CLINICAL TRIAL: NCT02220257
Title: Influence of Occurrence of Remission and Its Duration on Development of Chronic Complications of Type 1 Diabetes and Patient Outcome
Brief Title: The Influence of Partial Remission Phase of Type 1 Diabetes on Patient Outcome
Acronym: POZREM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Paweł Niedźwiecki, MD Paweł Niedźwiecki, Poznan University of Medical Sciences
Other Study IDs: REMISSIONDM1
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus Type 1; Remission of Type 1 Diabetes; Chronic Complications of Diabetes
Keywords: diabetes mellitus type 1; remission, honeymoon; microangiopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Newly diagnosed type 1 diabetes

SUMMARY:
Natural course of diabetes mellitus involves gradual reduction of β cell mass within islets of Langerhans in the pancreas. Symptoms of diabetes present when the mass of insulin-producing cells reaches a point where insulin concentration does not suffice to maintain proper glycaemia. In many patients β cells regenerate shortly after the diagnosis of diabetes and initiation of insulin therapy. This phenomenon is called a remission.

The aim of this study is to asses the influence of occurrence and duration of remission on development of chronic complications of diabetes and patients outcome.

DETAILED DESCRIPTION:
Natural course of diabetes mellitus involves gradual reduction of β cell mass within islets of Langerhans in the pancreas. Symptoms of diabetes present when the mass of insulin-producing cells reaches a point where insulin concentration does not suffice to maintain proper glycaemia. In many patients β cells regenerate shortly after the diagnosis of diabetes and initiation of insulin therapy. This phenomenon is called a remission.

The aim of this study is to asses influence of occurrence and duration of remission on development of chronic complications of diabetes and patients outcome.

Clinical remission was defined as time in which all of the following criteria were met: HbA1c below 6.5 % , dose of exogenous insulin below 0.3 U / kg body weight and serum C-peptide concentration above 0.5 ng / ml. Patients were divided into those who were in remission at any time during follow-up (remitters) and non-remitters.

At follow-up occurrence of chronic microvascular complications of diabetes (retinopathy, diabetic kidney disease and neuropathy) was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed type 1 diabetes according to ADA (American Diabetes Association) 1997 criteria.
2. Age 18-35 years
3. Education with regard to intensive functional insulin therapy at the time of diagnosis
4. Patient consent to participation in the study

Exclusion Criteria:

1. Acute inflammation (serum C-reactive protein concentration (hsCRP) >10mg/L, leukocytosis >15x109/L, erythrocyte sedimentation rate (OB) >30 mm/h)
2. Laboratory signs of liver damage: alanine and aspartate aminotransferase elevated 2-fold over the upper limit of normal range
3. History of other chronic diseases (e.g. asthma, neoplastic diseases, liver cirrhosis)
4. Other autoimmunological diseases other than diabetes
5. Not confirming type 1 diabetes after obtaining results of autoantibodies

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study included 240 consecutive patients, including 77 women and 143 men hospitalized at the Department of Internal Medicine and Diabetology of Poznan University of Medical Sciences between 2004 and 2007 due to newly diagnosed type 1 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Development of chronic complication of diabetes (retinopathy or neuropathy or nephropathy) | Evaluation for chronic complications of diabetes was conducted after a period of no less than 5 years from diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Niedźwiecki, MD, Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- Franciszek Raszeja Hospital; Poznan University of Medical Science, Poznan, Greater Poland Voivodeship, Poland